CLINICAL TRIAL: NCT00488345
Title: A Multicenter, Open-Label, Ascending Multiple-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Tigecycline in Patients 8 to 11 Years of Age With Selected Serious Infections
Brief Title: Study Evaluating the Pharmacokinetics (PK), Safety, and Tolerability of Tigecycline in Patients 8 to 11 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074K4-2207
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-09

CONDITIONS: Bacterial Infections; Intra-Abdominal Infection; Pneumonia, Bacterial; Skin Diseases, Bacterial; Skin Diseases, Infectious
Keywords: cIAI; cSSSI; CAP; Child
MeSH Terms: conditions — Bacterial Infections; Intraabdominal Infections; Pneumonia, Bacterial; Skin Diseases, Bacterial; Skin Diseases, Infectious | interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): 0.75 mg/kg (up to a maximum dose of 50 mg for each dose) of tigecycline every 12 hours infused over approximately 30 minutes. Escalation to next dose cohort will occur only after safety and tolerability at preceding dose have been established by sponsor (after tigecycline LDOT data are received) and if at least 5 of 6 PK samples per patient have been received by central laboratory in acceptable condition for 10 to 12 patients in cohort. Treatment period of tigecycline will be a minimum of 3 days (unless patient is considered a treatment failure before this time) and a maximum of 14 days. On or after Day 4, based on investigator's decision, patients can switch to oral antibiotic therapy (to be chosen and provided by the investigator) and discharged after collection of planned PK samples.
  Interventions: Drug: Tygacil
- B (Experimental): 1 mg/kg (up to a maximum dose of 50 mg for each dose) of tigecycline every 12 hours infused over approximately 30 minutes. Escalation to next dose cohort will occur only after safety and tolerability at preceding dose have been established by sponsor (after tigecycline LDOT data are received) and if at least 5 of 6 PK samples per patient have been received by the central laboratory in acceptable condition for 10 to 12 patients in the cohort. Treatment period of tigecycline will be a minimum of 3 days (unless the patient is considered a treatment failure before this time) and a maximum of 14 days. On or after Day 4, based on investigator's decision, patients can switch to oral antibiotic therapy (to be chosen and provided by the investigator) and discharged after collection of planned PK samples.
  Interventions: Drug: Tygacil
- C (Experimental): 1.25 mg/kg (up to maximum dose of 50 mg for each dose) of tigecycline every 12 hours infused over approximately 30 minutes. Treatment period of tigecycline will be a minimum of 3 days (unless patient is considered a treatment failure before this time) and a maximum of 14 days. On or after Day 4, based on investigator's decision, patients can switch to oral antibiotic therapy (to be chosen and provided by the investigator) and discharged after collection of planned PK samples.
  Interventions: Drug: Tygacil

INTERVENTIONS:
Drug: Tygacil

SUMMARY:
To determine the pharmacokinetic profile and to evaluate the safety and tolerability of ascending multiple doses of tigecycline in patients aged 8 to 11 years with selected serious infections; complicated intra-abdominal infections (cIAI), complicated skin and skin structure infections (cSSSI), or community-acquired pneumonia (CAP).

ELIGIBILITY:
Inclusion Criteria

* Male or female patients aged 8 to 11 years, inclusive, willing and able to complete all activities required for the study
* Have a diagnosis of a serious infection (cIAI, cSSSI or CAP) requiring hospitalization and administration of IV antibiotic therapy during greater than or equal to 5 days
* Other inclusion criteria apply.

Exclusion criteria

* Patients with any concomitant condition or taking any concomitant medication that, in the opinion of the investigator, could preclude an evaluation of safety or efficacy responses or make it unlikely that the anticipated course of therapy or follow-up assessment will be completed (e.g., life expectancy < 30 days).
* Pregnant or breastfeeding female patients and female patients of childbearing potential who are unable or unwilling to take adequate contraceptive precautions.
* Previous participation in this clinical trial.
* Receipt of any investigational drugs or devices (defined as lacking any regulatory agency's approval within 4 weeks before administration of the first dose of tigecycline).
* Endocarditis; presence of an artificial heart valve or infected device that will not be removed.
* Known or suspected hypersensitivity to tigecycline or other compounds related to this class of antibacterial agents (i.e., tetracyclines).
* Known or suspected P. aeruginosa infection.
* Patients receiving immunosuppressive therapy that, in the opinion of the investigator, would decrease the patient's ability to eradicate the infection, including the use of high-dose corticosteroid.
* Receipt of an organ or bone marrow transplant.
* Presence of any of the following laboratory findings: Neutropenia (absolute neutrophil count < 1 × 109/L [< 1000/mm3]) , AST or ALT > 10 × the ULN or bilirubin > 3 × ULN, unless isolated hyperbilirubinemia is directly related to the acute process (for patients with cIAI).
* Patients with any of the following conditions:

  * Cystic fibrosis.
  * Active tuberculosis.
  * Congenital immunodeficiency.
  * Meningitis.
  * Septic shock.
  * Osteomyelitis (suspected or evident).
  * Refractory shock syndrome in which hemodynamic parameters cannot be maintained despite adequate supportive therapy.
  * Confirmed malignancy with patient receiving an active course of chemotherapeutic agents.
  * Known or suspected infection with human immunodeficiency virus (HIV) or positive test result for HIV antibody.
  * Known or suspected concomitant bacterial or parasitic infection requiring systemic treatment.
* cSSSI patients, the presence of decubitus ulcers, necrotizing fasciitis, gas gangrene, or skeletal infection;
* CAP patients who have been hospitalized within 14 days before the onset of symptoms;
* CAP Patients: Presence of any of the following for patients with pneumonia:

  * Postobstructive pneumonia.
  * Pulmonary abscess.
  * Empyema.
  * Known or suspected pulmonary infection with Pneumocystis carinii.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (33):
- United States (18):
  - Long Beach, California
  - Oakland, California
  - Orange, California
  - San Diego, California
  - Tampa, Florida
  - Louisville, Kentucky
  - Flint, Michigan
  - Jackson, Mississippi
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
  - Richmond, Virginia
- Brussels, Belgium
- Guadalarajara Jalisco, Mexico
- South Africa (4):
  - Parow
  - Pretoria
  - Themba
  - Worcester
- Taipei, Taipei, Taiwan
- Ukraine (8):
  - Kyiv, Kyiv Oblast
  - Lviv, Lviv Oblast
  - Uzhhorod, Uzhorod
  - Vinnitsa, Vynnitsa
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Vinnitsa

REFERENCES:
- [Derived] Purdy J, Jouve S, Yan JL, Balter I, Dartois N, Cooper CA, Korth-Bradley J. Pharmacokinetics and safety profile of tigecycline in children aged 8 to 11 years with selected serious infections: a multicenter, open-label, ascending-dose study. Clin Ther. 2012 Feb;34(2):496-507.e1. doi: 10.1016/j.clinthera.2011.12.010. Epub 2012 Jan 16. PMID 22249106

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-nine participants were screened and enrolled in the study, and 58 participants received at least 1 dose of tigecycline.
Groups:
- Tigecycline 0.75 mg/kg: 0.75 milligram per kilogram (mg/kg) intravenous (IV) infusion every 12 hours
- Tigecycline 1 mg/kg: 1 milligram per kilogram (mg/kg) IV infusion every 12 hours
- Tigecycline 1.25 mg/kg: 1.25 milligram per kilogram (mg/kg) IV infusion every 12 hours
Period: Overall Study
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Started | 17 | 21 | 20
Completed | 17 | 17 | 17
Not Completed | 0 | 4 | 3
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Unable to administer antibiotics at home | 0 | 1 | 0
Not completed — Institutional Review Board review | 0 | 0 | 1
Not completed — Surgical team recommendation | 0 | 1 | 0
Not completed — Parent/legal guardian request | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg | Total
Number analyzed (Participants) | 17 | 21 | 20 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 10.21 (1.15) | 10.20 (1.06) | 9.72 (0.94) | 10.04 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 8 | 27
  Male | 8 | 11 | 12 | 31
Selected Serious Infections [Number; unit: participants]
  Community Acquired Pneumonia | 7 | 8 | 4 | 19
  Complicated Intra-abdominal Infection | 6 | 6 | 12 | 24
  Complicated Skin and Skin Structure Infection | 4 | 7 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax: tigecycline serum concentration measured in nanograms per milliliter (ng/mL) determined by a validated liquid chromatography with mass spectrophotometric (LC/MS/MS) detection method. Peak concentration was taken directly from the observed data.
Time Frame: Day 3 (immediately post-dose, 0.75, and 2 hours post-dose)
Population: Modified intent to treat (mITT) population: participants who were screened, assigned to study medication and received at least one dose of study medication. N = number of participants with evaluable tigecycline concentration data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Number analyzed (Participants) | 17 | 19 | 16
ng/mL | 456 (347) | 1515 (1457) | 2599 (3643)

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Time of peak concentration taken directly from the observed data.
Time Frame: Day 3 (immediately post-dose, 0.75, and 2 hours post-dose)
Population: mITT; N = number of participants with evaluable tigecycline concentration data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Number analyzed (Participants) | 17 | 19 | 16
hours | 0.6 (0.2) | 0.5 (0.1) | 0.8 (0.6)

3. Primary Outcome: Area Under the Curve (AUCτ) From Time Zero to Time of Estimated Concentration at 12 Hours
Description: AUCτ: AUC between doses from time zero to the time of estimated concentration at 12 hours reported in nanograms * hours divided by milliliters (ng*h/mL) was calculated using the log-trapezoidal rule for decreasing concentrations and the linear-trapezoidal rule for increasing concentrations estimating the 12 hour drug concentration if necessary.
Time Frame: Day 3 (just before and immediately after infusion, and 0.75, 2, and 6 hours post-dose)
Population: mITT; N = number of participants with sufficient reported tigecycline concentration data to estimate AUC.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Number analyzed (Participants) | 16 | 18 | 13
ng*h/mL | 1650 (529) | 2557 (1196) | 3196 (1704)

4. Primary Outcome: Weight Normalized Drug Clearance (CLW)
Description: Weight normalized drug clearance measured in liters per hour per kilogram (L/hr/kg). Drug clearance (CL) was determined as the ratio of dose/area under the concentration-time curve from time zero (start of infusion) to 12 hours (start of next infusion) (AUCτ). CLW was determined as the ratio of CL/weight.
Time Frame: Day 3 (just before and immediately after infusion, and 0.75, 2, and 6 hours post-dose)
Population: mITT; N = number of participants with sufficient reported tigecycline concentration data to estimate AUC.
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Number analyzed (Participants) | 16 | 18 | 13
L/hr/kg | 0.490 (0.130) | 0.498 (0.335) | 0.528 (0.384)

5. Secondary Outcome: Population Pharmacokinetic (PK) Model: Volume of Distribution
Description: Two compartment model with linear clearance and effect of weight on clearance using pooled PK data from 2 pediatric studies. All concentration-time data were combined and analyzed using population PK methods to investigate potential influence of age, weight, and height (dose, tigecycline concentrations, times, subject weight, height, age, body surface area, serum creatinine, estimated creatinine clearance, serum bilirubin.
Time Frame: 3074K4-2207: Day 3 just before and immediately after infusion, and 0.75, 2, and 6 hours post-dose; 3074A1-110: just before and 0.5, 0.75, 1, 2, 3, 4, 8, 12, 24, 36, and 48 hours after start of infusion
Population: Separate population pharmacokinetic analysis results are not available for the current study as more than 1 study was involved in this analysis based on pooled data from pediatric studies 3074A1-110 and 3074K4-2207.
Groups:
- Tigecycline 0.75 mg/kg, 1 mg/kg, 1.25 mg/kg: 0.75, 1 mg/kg, and 1.25 milligram per kilogram (mg/kg) intravenous (IV) infusions every 12 hours
Arm/Group | Tigecycline 0.75 mg/kg, 1 mg/kg, 1.25 mg/kg
Number analyzed (Participants) | 0

6. Primary Outcome: Percentage of Participants With Clinical Response (CR) to Tigecycline at Last Day of Therapy (LDOT) and Test-of-Cure (TOC) Assessment
Description: CR = Cure: resolution of all signs, symptoms (SS) of infection (INF) or improvement, no further antibacterial therapy (AT) necessary; Improved (IMP): SS IMP to extent that switch to oral AT deemed appropriate; Failure: lack of response, required additional AT, initial recovery then deterioration requiring further AT, death due to the INF after day 2, death due to treatment (TR)-related adverse event (AE), required non-routine surgical TR >48 hours after 1st dose of TR due to failure to IMP or clinical worsening. TOC = CR, vital signs, physical exam, laboratory results, concomitant TR, and AEs.
Time Frame: Day 14 or LDOT, TOC Visit (10 to 21 days after last dose of total antibiotic therapy)
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Number analyzed (Participants) | 17 | 21 | 20
percentage of participants
  Cure: LDOT | 82.4 | 52.4 | 30.0
  Improved: LDOT | 17.6 | 28.6 | 55.0
  Failure: LDOT | 0.0 | 0.0 | 0.0
  Indeterminate: LDOT | 0.0 | 19.0 | 15.0
  Cure: TOC | 94.1 | 76.2 | 75.0
  Failure: TOC | 5.9 | 4.8 | 10.0
  Indeterminate: TOC | 0.0 | 19.0 | 15.0

7. Secondary Outcome: Population Pharmacokinetic (PK) Model: Clearance
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Arm/Group | Tigecycline 0.75 mg/kg, 1 mg/kg, 1.25 mg/kg
Number analyzed (Participants) | 0

8. Secondary Outcome: Population Pharmacokinetic (PK) Model: Effect of Weight
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Arm/Group | Tigecycline 0.75 mg/kg, 1 mg/kg, 1.25 mg/kg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: mITT population. An Adverse Event(AE) term may be reported as both a serious and a non-serious AE, but are distinct events. AE may = serious for one subject and non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Tigecycline 0.75 mg/kg | Tigecycline 1 mg/kg | Tigecycline 1.25 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/21 | 1/20
Other Adverse Events (participants affected / at risk) | 11/17 | 16/21 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline 0.75 mg/kg (N=17) | Tigecycline 1 mg/kg (N=21) | Tigecycline 1.25 mg/kg (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline 0.75 mg/kg (N=17) | Tigecycline 1 mg/kg (N=21) | Tigecycline 1.25 mg/kg (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 13 | 12
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 11 | 11
Asthenia (General disorders) | 0 | 1 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0
Crepitations (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medical device pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood amylase increased (Investigations) | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 2 | 2
Platelet count increased (Investigations) | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.